CLINICAL TRIAL: NCT05078424
Title: A Randomized Controlled Trial of Cognitive Behavioural Therapy for Youths With Depressive and Anxiety Symptoms in Hong Kong
Brief Title: Cognitive Behavioural Therapy for Youths With Depressive and Anxiety Symptoms in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Federation of Youth's Group (HKFYG) (Other); Hong Kong Playground Association (Unknown); Hong Kong Children and Youth Services (Unknown); St. James' Settlement (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chair Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LevelMind@JC CBT
Record Dates: First submitted 2021-09-06; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
Keywords: Randomized Controlled Trial; Cognitive Behavioural Therapy; Youths; Depressive and Anxiety Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Treatment group (Experimental): This group receives CBT interventions that aim to improve mental well-being, depressive and anxiety symptoms in young people.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Wait-list Control group (No Intervention): This group does not receive CBT intervention but will receive appropriate intervention after the CBT treatment group and follow-up phases complete.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — CBT is a well-established, evidence-based intervention frequently used for easing depressive and anxiety symptoms. The intervention will be delivered for 6-7 sessions, each session lasts for 1.5 hours, in the format of a group for a period of 6-7 weeks by frontline social or youth workers trained by professional CBT clinicians. Core treatment components include mood monitoring, emotion education, behavioural activation, emotion cycle/ ABC model, identification of automatic thoughts, and cognitive restructuring. It is designed to improve youths' abilities/ skills in handling their moods to have better emotional management.
  Arms: CBT Treatment group

SUMMARY:
The proposed study is a randomized controlled trial (RCT) that aims to examine the effectiveness of cognitive behavioural therapy in reducing depressive and anxiety symptoms for youths in Hong Kong. It is to be carried out with 120 youths aged 12 - 24 recruited from a series of community-based LevelMind@JC hubs, funded by the Hong Kong Jockey Club Charities Trust. It is designed to improve the youths' abilities/ skills in handling moods to have better emotional management. A written informed consent will be signed by participants. Researchers will perform cognitive behavioural therapy on youths who agree to join the study.

ELIGIBILITY:
Inclusion Criteria:

* LevelMind@JC users with mild to moderate distress level (n=120);
* have sufficient proficiency in Chinese to understand verbal instructions and give informed consent;

Exclusion Criteria:

* known diagnosis of intellectual disability
* organic brain disorder
* photosensitive epilepsy
* significant visual, auditory or balance impairment
* current or previous use of illicit drugs
* known psychiatric diagnosis (stabilized diagnosis and treatment)
* receiving any psychosocial treatment for social withdrawal such as CBT or;
* current or active suicidal ideation or attempts.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in depressive and anxiety levels | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Depression Anxiety Stress Scales (DASS), scores ranging from 0-42 for each subscale, with higher scores representing worse outcome
Change in social anxiety levels | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Social Interaction Anxiety Scale (SIAS), scores ranging from 0-80 with higher scores representing higher levels of social anxiety hence worse outcome
Change in depressive levels | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Patient Health Questionnaire-9 (PHQ-9), scores ranging from 0-27 with higher scores representing higher depressive levels hence worse outcome
Change in distress levels | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Kessler Psychological Distress Scale (K6), scores ranging from 0-25 with higher scores representing higher distress hence worse outcome
Change in depressive symptoms | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Beck Depression Inventory II (BDI-II), scores ranging from 0-63 with higher scores representing severe depressive symptoms hence worse outcome
Change in anxiety symptoms | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Beck Anxiety Inventory (BAI), scores ranging from 0-36 with higher scores representing severe anxiety symptoms hence worse outcome
Change in anxiety levels | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Generalized Anxiety Stress Scale-7 (GAD-7), scores ranging from 0-21 with higher scores representing higher anxiety levels hence worse outcome

SECONDARY OUTCOMES:
Change in functioning | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Role Functioning Scale (RFS), scores ranging from 1-28 with higher scores representing better functioning
Change in social and occupational functioning | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Social and Occupational Functioning Assessment Scale (SOFAS), scores ranging from 0-100 with higher scores representing better functioning
Change in quality of life | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  12-item Short Form Survey (SF-12), scores ranging from 0-100 with higher scores representing better quality of life
Change in self-harm | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Self-harming behaviour, plans and thoughts, recording as binary response (0=No, 1=Yes)
Change in resilience | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Connor-Davidson Resilience Scale (CD-RISC), scores ranging from 0-100 with higher scores indicating higher resilience
Change in future outlook | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Future Outlook Inventory (FOI), scores ranging from 1-70 with higher scores indicating greater degree of future consideration
Change in self-esteem | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Rosenberg Self Esteem Scale (RSE), scores ranging from 0-30 with higher scores indicating higher self-esteem
Change in mindfulness | Baseline, after 7 weeks of intervention/wait, and 1 month after post-intervention
  Mindful Attention Awareness Scale (MAAS), scores ranging from 1-6 with higher scores indicating higher mindful awareness

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No